CLINICAL TRIAL: NCT01705509
Title: The Effects of Ranolazine on CPET Parameters in Ischemic Cardiomyopathy Patients (ERIC)
Acronym: ERIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to lack of resources.
Sponsor: Cardiovascular Institute of the South Clinical Research Corporation (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20121250
Record Dates: First submitted 2012-10-10; First posted 2012-10-12 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Cardiomyopathy
Keywords: The Effects of Ranolazine on CPET Parameters in Ischemic; Cardiomyopathy Patients
MeSH Terms: conditions — Cardiomyopathies | interventions — Ranolazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ranolazine Treatment Arm (Other): All patients who meet the criteria of ischemia will receive ranolazine after enrollment. The initial CPET will serve as the control. The second CPET after 30-days of therapy will serve as the therapy arm. CPET parameters will be assessed and compared both on and off therapy.
  Interventions: Drug: Ranolazine

INTERVENTIONS:
Drug: Ranolazine — The intervention will be ranolazine therapy after the initial CPET. The initial CPET will identify patients with underlying ischemia and serve as a baseline study. Patients whose CPET results meet the criteria for ischemia will be started on Ranexa 500mg BID and advanced within one week +/-4 days to 1000mg BID. A second CPET will be performed after 4 weeks +/- 4 days of maximum therapy. CPET results before and after therapy will undergo a statistical comparison. The initial off treatment CPET measurement will serve as the control to assess changes found during therapy.
  Other Names: Ranexa

SUMMARY:
This is a proof of concept trial using ranolazine, a medication, in patients with known Coronary Artery Disease and reduced left ventricular function, EF < 40%. We propose that ranolazine therapy will result in demonstrative improvements in cardiac function that can be objectively assessed using the parameters measured with CPET. We propose that demonstrative improvement in CPET parameters on ranolazine will translate into improved patient outcomes for this patient population.

DETAILED DESCRIPTION:
Selected patients will undergo a CPET evaluation. The initial CPET will identify patients with underlying ischemia and serve as a baseline study. Ischemia will be assessed using: 1) peak VO2: measures the peak transport of O2 to the tissues when O2 extraction from the blood is maximal; 2) the anaerobic threshold (AT): measures the sustainable work capacity in units of VO2; 3) the O2-pulse measurements at the AT peak VO2: estimate stroke volume at those levels of exercise; and 4) the relationship of O2 uptake to work rate (ΔVO2/ΔWR): provides information on the ability of the cardiac output to increase. Patients whoseCPET results meet the criteria for ischemia will be started on Ranexa 500mg BID and advanced within one week +/-4 days to 1000mg BID. A second CPET will be performed after 4 weeks +/- 4 days of maximum therapy. CPET results before and after therapy will undergo a statistical comparison. The initial off treatment CPET measurement will serve as the control to assess changes found during therapy. No medication changes or revascularization procedures will occur during the study. If patients require and undergo a medication change or a revascularization procedure, they will be excluded from the study.

Patients will be contacted at the completion of week one prior to up titration, then at the end of week two to ensure tolerance and compliance with the 1000mg BID dose. Patients will perform the second CPET study at week four +/- 1 week. The trial medication will be assessed and counted to ensure that patients have taken there allotted pill count for the duration of the study. Patients who are found to be noncompliant of less than 80% will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age will be enrolled in the trial.
* Stable patients without hospitalizations, medication changes or cardiac intervention within one month of the study will be enrolled.
* Patients must be able to complete the CPET protocol and must have demonstrable ischemia on the initial CPET evaluation.
* Patients must have a documented ejection fraction < 40%

  a. LV function can be assessed via: i. Echocardiogram ii. MUGA or Nuclear Perfusion Scan iii. Left ventriculogram
* Patients must be Ranexa naive and without contraindication for Ranexa therapy.

Exclusion Criteria:

* QTc>500 msec on resting EKG
* Hepatic Impairment (Child-Pugh class A, B or C)
* Have received prior treatment with ranolazine
* Treatment with QT prolonging drugs as class 1A (e.g., quinidine), class III (e.g., sotalol, dofetilide) anti-arrhythmics, amiodarone and anti-psychotics (e.g., thioridazine, ziprasidone)
* Treatment with potent or moderately potent CYP3A inhibitors including ketoconazole and other azole antifungals, diltiazem, verapamil, macrolide antibiotics, HIV protease inhibitors or consumption of grapefruit juice or grapefruit juice containing products
* Have participated in another trial of an investigational device or drug within 30 days of screening
* Have end stage renal disease requiring dialysis
* Have any chronic illness likely to effect compliance with the protocol
* Have second or third degree atrioventricular block in the absence of a functioning ventricular pacemaker
* Have uncontrolled clinically significant cardiac arrhythmias, or a history of ventricular fibrillation, torsade de pointes, or other life-threatening ventricular arrhythmias
* Uncontrolled HTN defined as BP > /= 160/100 mm Hg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Agostino G Ingraldi, M.D., Principal Investigator — Cardiovascular Institute of the South
Locations (1):
- Cardiovascular Institute of the South, Lafayette, Louisiana, United States

REFERENCES:
- [Background] Lloyd-Jones D, Adams RJ, Brown TM, Carnethon M, Dai S, De Simone G, Ferguson TB, Ford E, Furie K, Gillespie C, Go A, Greenlund K, Haase N, Hailpern S, Ho PM, Howard V, Kissela B, Kittner S, Lackland D, Lisabeth L, Marelli A, McDermott MM, Meigs J, Mozaffarian D, Mussolino M, Nichol G, Roger VL, Rosamond W, Sacco R, Sorlie P, Stafford R, Thom T, Wasserthiel-Smoller S, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2010 update: a report from the American Heart Association. Circulation. 2010 Feb 23;121(7):948-54. doi: 10.1161/CIRCULATIONAHA.109.192666. No abstract available. PMID 20177011
- [Background] McMurray JJ, Petrie MC, Murdoch DR, Davie AP. Clinical epidemiology of heart failure: public and private health burden. Eur Heart J. 1998 Dec;19 Suppl P:P9-16. PMID 9886707
- [Background] Wenger NK, Chaitman B, Vetrovec GW. Gender comparison of efficacy and safety of ranolazine for chronic angina pectoris in four randomized clinical trials. Am J Cardiol. 2007 Jan 1;99(1):11-8. doi: 10.1016/j.amjcard.2006.07.052. Epub 2006 Nov 2. PMID 17196454
- [Background] Belardinelli L, Shryock JC, Fraser H. Inhibition of the late sodium current as a potential cardioprotective principle: effects of the late sodium current inhibitor ranolazine. Heart. 2006 Jul;92 Suppl 4(Suppl 4):iv6-iv14. doi: 10.1136/hrt.2005.078790. PMID 16775092
- [Background] Chaitman BR. Ranolazine for the treatment of chronic angina and potential use in other cardiovascular conditions. Circulation. 2006 May 23;113(20):2462-72. doi: 10.1161/CIRCULATIONAHA.105.597500. No abstract available. PMID 16717165
- [Background] Belardinelli R, Lacalaprice F, Carle F, Minnucci A, Cianci G, Perna G, D'Eusanio G. Exercise-induced myocardial ischaemia detected by cardiopulmonary exercise testing. Eur Heart J. 2003 Jul;24(14):1304-13. doi: 10.1016/s0195-668x(03)00210-0. PMID 12871687
- [Background] Contini M, Andreini D, Agostoni P. Cardiopulmonary exercise test evidence of isolated right coronary artery disease. Int J Cardiol. 2006 Nov 10;113(2):281-2. doi: 10.1016/j.ijcard.2005.09.033. Epub 2005 Nov 28. PMID 16316693
- [Background] Klainman E, Fink G, Lebzelter J, Zafrir N. Assessment of functional results after percutaneous transluminal coronary angioplasty by cardiopulmonary exercise test. Cardiology. 1998 May;89(4):257-62. doi: 10.1159/000006797. PMID 9643272
- [Background] Itoh, H et al. Oxygen uptake abnormalities during exercise in coronary artery disease. In Cardiopulmonary Exercise Testing and Cardiovascular Health. Edited by K. Wasserman, Published by Futura Publishing Company, Armonk NY, 2002.

RESULTS

PARTICIPANT FLOW:
Groups:
- CPET Control / CPET With Ranexa: The initial CPET will identify patients with underlying ischemia and serve as a baseline study. Patients whose CPET results meet the criteria for ischemia will be started on Ranexa 500mg BID and advanced within one week +/-4 days to 1000mg BID. A second CPET will be performed after 4 weeks +/- 4 days of maximum therapy. CPET results before and after therapy will undergo a statistical comparison.
Period: Inclusion CPET
Arm/Group | CPET Control / CPET With Ranexa
Started | 14
Completed | 7
Not Completed | 7
Not completed — Screen Failure | 5
Not completed — Withdrawal by Subject | 2
Period: CPET w/ Ranexa
Arm/Group | CPET Control / CPET With Ranexa
Started | 7
Completed | 5
Not Completed | 2
Not completed — Screen Failure | 2

BASELINE CHARACTERISTICS:
Groups:
- CPET Control / CPET With Ranexa: Enrolled patients will undergo a CPET evaluation. Beta Blockers will be held day prior to and day of CPET. The initial CPET will identify patients with underlying ischemia and serve as a baseline study. Patients whose CPET results meet the criteria for ischemia will be started on Ranexa 500mg B ID and advanced within one week +/-4 days to 1000mg BID. A second CPET will be performed after 4 weeks +/- 4 days of maximum therapy. CPET results before and after therapy will undergo a statistical comparison. The initial off treatment CPET measurement will serve as the control to assess changes found during therapy. No medication changes or revascularization procedures will occur during the study.
Arm/Group | CPET Control / CPET With Ranexa
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 9
Age, Continuous [Mean (Full Range); unit: years] | 68 [58 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Cardiopulmonary Exercise Test Parameters (CPET).
Description: CPET parameters assessed will include the peak VO2: measures the peak transport of O2 to the tissues when O2 extraction from the blood is maximal; 2) the anaerobic threshold (AT): measures the sustainable work capacity in units of VO2; 3) the O2-pulse measurements at the AT and peak VO2: estimate stroke volume at those levels of exercise; and 4) the relationship of O2 uptake to work rate (ΔVO2/ΔWR): provides information on the ability of the cardiac output to increase.
Time Frame: 30 days
Population: Number of Participants who Reached CPET Milestones
Measure: Count of Participants; unit: Participants
Groups:
- Control: All patients who meet the criteria of ischemia will receive ranolazine after enrollment. The initial CPET will serve as the control. The second CPET after 30-days of therapy will serve as the therapy arm. CPET parameters will be assessed and compared both on and off therapy.
  Ranolazine: The intervention will be ranolazine therapy after the initial CPET. The initial CPET will identify patients with underlying ischemia and serve as a baseline study. Patients whose CPET results meet the criteria for ischemia will be started on Ranexa 500mg BID and advanced within one week +/-4 days to 1000mg BID. A second CPET will be performed after 4 weeks +/- 4 days of maximum therapy. CPET results before and after therapy will undergo a statistical comparison. The initial off treatment CPET measurement will serve as the control to assess changes found during therapy.
Arm/Group | Control
Number analyzed (Participants) | 14
Participants
  Failed Initial CPET | 5
  Withdrew Prior to CPET | 2
  Screenfailed due to Ranolazine Intolerance | 2
  Completed | 5

ADVERSE EVENTS:
Time Frame: 30 days.
Groups:
- CPET Control / CPET With Ranexa: The initial CPET will identify patients with underlying ischemia and serve as a baseline study. Patients whose CPET results meet the criteria for ischemia will be started on Ranexa 500mg BID and advanced within one week +/-4 days to 1000mg BID. A second CPET will be performed after 4 weeks +/- 4 days of maximum therapy.
Arm/Group | CPET Control / CPET With Ranexa
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 4/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPET Control / CPET With Ranexa (N=14)
CAD (Ranexa 1000mg BID Treatment) (Cardiac disorders) | 1 (1) — Coronary artery disease
Ranexa Intolerant (Ranexa 1000mg BID Treatment) (General disorders) | 2 (2) — Subject intolerant to Ranexa.
Headache (Ranexa 1000mg BID Treatment) (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2012-09-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT01705509/ICF_000.pdf
  • Study Protocol (2013-02-24): https://cdn.clinicaltrials.gov/large-docs/09/NCT01705509/Prot_001.pdf